CLINICAL TRIAL: NCT06470672
Title: A Phase 2 Study of SHR-A1921 Combined Adebrelimab in Endocrine Therapy-failed HR-positive, HER2-negative Advanced Breast Cancer
Brief Title: Study of SHR-A1921 Combined Adebrelimab in HR-positive, HER2-negative Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Hongxia Wang, Chief Physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-MUL-IIT-SHRA1921-SHR1316
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-06

CONDITIONS: Advanced Breast Cancer; Hormone-receptor-positive Breast Cancer; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SHR-A1921+Adebrelimab (Experimental): Via intravenous infusion
  Interventions: Drug: SHR-A1921; Drug: Adebrelimab

INTERVENTIONS:
Drug: SHR-A1921 — Anti-TROP-2 ADC
Drug: Adebrelimab — PD-L1 inhibitor

SUMMARY:
Our study is aimed to evaluate the efficacy and safety of novel ADC named SHR-A1921 combined with Adebrelimab in endocrine therapy-failed HR (Hormone Receptor)-positive, HER2-negative advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 75 years old, female patients with breast cancer;
* ECOG PS Score: 0~1;
* Histologically or cytologically confirmed HR-positive, HER2-negative advanced or metastatic breast cancer;
* PD-L1 positive;
* Disease progression after at least prior 2 lines of endocrine therapy, and unable to benefit from further endocrine therapy determined by investigator, of which at least one line of CDK4/6 inhibitor-based treatment; if recurrence or metastasis within 2 years after completion of adjuvant endocrine therapy, marked as first-line treatment;
* Prior at least 1 line of systemic chemotherapy in recurrent or metastatic setting;
* Based on RECIST v1.1, at least one measurable lesion;
* Patients must have a life expectancy ≥ 3 months;
* Adequate organ function and marrow function (no corrective treatment within 14 days before first dose);
* Women of childbearing potential (WOCBP) should agree to use an effective method of contraception and no lactation from the initiation of screening to 7 months after the last dose of study therapy; WOCBP should have a negative serum pregnancy result within 7 days before the first dose of study therapy;
* Willing and able to provide written informed consent and comply with the requirements and restrictions in the protocol.

Exclusion Criteria:

* Has leptomeningeal metastasis confirmed by MRI or lumbar puncture;
* Has CNS metastasis confirmed by radiology, except following conditions: ①asymptomatic brain metastasis that is not required to radiotherapy or surgery immediately; ②prior local therapy (e.g. radiotherapy or surgery) for brain or dural metastasis, of which stable disease lasting at least 4 weeks confirmed by radiography, and symptomatic therapy (e.g. hormone, mannitol, bevacizumab) has been stopped beyond 2 weeks with no clinical symptom;
* Prior anti-TROP-2 treatment;
* Has received or been receiving PD-(L)1 inhibitors and/or ADC containing a topoisomerase inhibitor-like payload;
* Existence of third space fluid (e.g. massive ascites, pleural effusion, pericardial effusion) that is not well controlled by effective methods, e.g. drainage;
* Has received antitumor surgery, radiotherapy, chemotherapy, targeted therapy or immunological therapy within 4 weeks before first dose of study therapy; has received antitumor endocrine therapy within one week before first dose of study therapy;
* Use of other antitumor systemic treatment during the study;
* Has active autoimmune disease or a history of autoimmune disease;
* Known history of immunodeficiency, including HIV-positive, other acquired or innate immunodeficient disease, or known history of organ transplantation;
* Has active hepatitis B (HBsAg-positive and HBV DNA≥500 IU/mL), hepatitis C (positive for HCV antibody and HCV RNA above ULN) and hepatic cirrhosis;
* Has an active infection requiring antibiotics, antiviral or antifungal treatment, or pyrexia >38.5℃ of unknown origin during the screening period before first dose of study therapy (patients with pyrexia due to cancer could be enrolled determined by investigator);
* Receiving immunosuppressive medication, or systemic corticosteroid therapy for the purpose of immunosuppression (prednisone at >10mg/d or equivalent dose of other corticosteroids), and continuous use within 2 weeks before the first dose of study therapy;
* Other malignancy within prior 5 years unless curatively treated with no evidence of disease for at least recent 3 years, except: curatively treated in situ cancer of the cervix, skin basal cell carcinoma or skin squamous cell carcinoma;
* Hypersensitivity to study therapy or any of its excipients;
* Has known clinically significant lung disease, including but not limited to: interstitial lung disease, pneumonitis, pulmonary fibrosis;
* Known history of uncontrolled cardiovascular clinical symptom or disease that is not well controlled;
* Has received a live vaccine within 4 weeks before first dose of study therapy, or potential to receive a live vaccine during the trial treatment;
* Other conditions that might influence the study and analysis of results in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
ORR by investigator | At baseline, at the time point of every 6 weeks, up to 2 years
  ORR (Objective response rate) is the percentage of evaluable patients with a confirmed investigator-assessed response of CR (complete response) or PR (partial response) per RECIST v1.1.

SECONDARY OUTCOMES:
DCR by investigator | At baseline, at the time point of every 6 weeks, up to 2 years
  DCR (Disease control rate) is the percentage of evaluable patients with a confirmed investigator-assessed response of CR (complete response), PR (partial response) or SD (stable disease) per RECIST v1.1.
DoR (Duration of Response) | Up to 2 years
  DoR is the time from the date of first detection of objective response (which is subsequently confirmed) until the date of objective radiographic disease progression.
PFS (Progression-Free Survival) | Up to 2 years
  PFS is the time from the date of first dose until the date of objective radiographic disease progression or death (by any cause in the absence of progression).
OS (Overall Survival) | Up to 2 years
  OS is the time from the date of first dose until the date of death by any cause.
Safety (incidence rate of adverse event) | From time of informed consent provided to 3 months after the last dose of study therapy
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. Percentage of participants who experienced an adverse event and discontinued study drug due to an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Wang, Principal Investigator — Fudan Cancer Hospital
Locations (1):
- Fudan Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No